CLINICAL TRIAL: NCT00841256
Title: ... Study to Evaluate Efficacy and Safety of Perennial Sublingual SIT With a Solution of Grass Pollen Allergen ... in Children With Clinically Relevant Grass Pollen Sensitivity in Comparison to a ... Standard Treatment With Add on Placebo
Brief Title: Multicenter Trial of Sublingual Immunotherapy With a Solution of Grass Pollen Allergen Extract in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL0506st; 2006-005911-82 (EudraCT Number)
Record Dates: First submitted 2008-04-22; First posted 2009-02-11 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: specific immunotherapy; SIT; SLIT; sublingual

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immunotherapy (Experimental): Grass pollen allergens in a water/glycerol solution
  Interventions: Biological: Grass pollen allergens in a water/glycerol solution
- Placebo (Placebo Comparator): Water/glycerol solution with phosphate buffered saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Grass pollen allergens in a water/glycerol solution — In total up to 4 drops (dose for maintenance therapy) are administered under the tongue.
  Other Names: Allerslit forte grasses
  Arms: Immunotherapy
Drug: Placebo — Placebo was given in the same way as the sublingual active treatment. Symptomatic standard treatment, i.e. antihistamines and glucocorticoids as well as alphamimetics is allowed during grass pollen season.
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
Evaluation of safety and efficacy of sublingual immunotherapy with grass pollen allergens formulated as solution in comparison to a symptomatic standard treatment with add on placebo in grass pollen allergic children suffering from allergic rhinitis/rhinoconjunctivitis with or without bronchial asthma.

DETAILED DESCRIPTION:
Although highly effective, subcutaneous administration of allergens may cause inconvenience in some patients. Alternative routes, e.g. nasal and oral, have therefore been investigated to find an immunotherapy regimen largely accepted by all groups of patients, including children.

Sublingual specific immunotherapy (SLIT) may represent a more acceptable route of immunotherapy. It may be an optimal therapy option especially for children because they often fear injections.

In this study children are to be treated with a preparation of a grass pollen allergen extract in a water/glycerol solution with phosphate buffered saline in comparison to a symptomatic standard treatment with add on placebo, in order to investigate efficacy and safety of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* 4 - <12 years (at the time of inclusion)
* Positive SPT
* Positive EAST
* Positive CPT

Exclusion Criteria:

* Serious chronic diseases
* Other perennial allergies

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 207 (Actual)
Dates: Start 2008-02; Primary Completion 2012-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Changes of Symptom-Medication-Score | After 1 year of treatment
  The change of the area under the curve of the symptom and medication score (SMS) from the baseline season to the season after 1 year of treatment.

SECONDARY OUTCOMES:
Evaluation of the documentation of adverse events (AEs) | Entire treatment period
  Safety of treatments during the entire treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Wahn, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Klinik für Paediatrie Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Result] Wahn U, Klimek L, Ploszczuk A, Adelt T, Sandner B, Trebas-Pietras E, Eberle P, Bufe A; SLIT Study Group. High-dose sublingual immunotherapy with single-dose aqueous grass pollen extract in children is effective and safe: a double-blind, placebo-controlled study. J Allergy Clin Immunol. 2012 Oct;130(4):886-93.e5. doi: 10.1016/j.jaci.2012.06.047. Epub 2012 Aug 29. PMID 22939758
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de
- See also: Click here for information about this trial in the European Clinical Trials Register — https://www.clinicaltrialsregister.eu/ctr-search/trial/2006-005911-82/DE